CLINICAL TRIAL: NCT04357132
Title: Functional Response to Immersive Virtual Reality in Pediatric Patients Post-Laparoscopic Appedectomy
Brief Title: Virtual Reality for Appendectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-0258
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Appendix Rupture; Pain; Pain, Postoperative
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: 60 participants assigned to one of two groups. VR- Distraction and VR-Biofeedback
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Biofeedback (Other)
  Interventions: Other: VR-Biofeedback
- VR-Distraction (Other)
  Interventions: Other: VR-Distraction

INTERVENTIONS:
Other: VR-Biofeedback — Participants will be instructed to use the Mindful Aurora Application
  Arms: VR-Biofeedback
Other: VR-Distraction — Participants will be instructed to use one of four applications
  Arms: VR-Distraction

SUMMARY:
To determine the impact of VR-Biofeedback and VR-Distraction on pain and medication utilization in children and adolescents undergoing surgery for ruptured appendix.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 - 18 years
* Able to read, understand, and speak English
* Patients in the immediate postoperative period following laparoscopic appendectomy for ruptured appendix

Exclusion Criteria:

* Outside of age range (<8 or >18 years)
* History of developmental delays, uncontrolled psychiatric conditions, or neurological conditions (especially epilepsy and/or significant motion sickness/nausea/vomiting)
* History of vertigo, dizziness, and/or seizure disorders
* Conditions that would preclude the application of the VR headset, such as craniofacial deformities
* History of chronic pain, frequent opioid use and/or active cancer therapy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Effect on VR-biofeedback on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a visual analog scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect on VR-biofeedback on anxiety | Immediately after VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect on VR-biofeedback on anxiety | 15 minutes after VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect on VR-biofeedback on anxiety | 30 minutes after VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect of VR-biofeedback on pain | Postoperatively 24 - 90 hours.
  Pain scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Effect of VR-biofeedback on medication use | 24-90 hours
  Amount of pain medications used will be collected
Effect of VR-distraction on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect of VR-distraction on anxiety | Immediately after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect of VR-distraction on anxiety | 15 minutes after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect of VR-distraction on anxiety | 30 minutes after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect of VR-distraction on pain | Postoperatively 24 - 90 hours.
  Pain scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Effect of VR-distraction on medication use | 24-90 hours
  Pain medications used will be collected

SECONDARY OUTCOMES:
Role of anxiety on changes in pain | One time prior to study visit
  Participants will complete a questionnaire regarding anxiety
Role of pain catastrophizing | One time prior to study visit
  Participants will complete a questionnaire regarding pain

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Olbrecht, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States